CLINICAL TRIAL: NCT06231628
Title: Immediate and Short-term Outcomes of Imaging Guided Percutaneous Cementoplasty for Pelvic Bone Metastases
Brief Title: Imaging Guided Cementoplasty for Pelvic Bone Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Hosam Hasan Ali, Resident Radiology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maha Hosam
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Imaging Guided; Percutaneous Cementoplasty; Pelvic Bone Metstasis
Keywords: cementoplasty; metastasis; percutaneous; pelvis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cementoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): A single arm with patients with advanced cancer who have all of the following:
  1. refractory pain and/or gait disturbance caused by pelvic bone metastasis, did not respond to conservative treatment.
  2. osteolytic lesion (in predominance) suitable for the pain.
  3. limited life expectancy (less than 3 years) or stopping medical treatment.
  Exclusion criteria:
  There are no absolute contraindications for the procedure; however, the relative contraindications are:
  1. patients in poor condition with an expected survival period of less than 3 months.
  2. patients with stable course, with long life expectancy (more than 3 years) or those considered candidates for major pelvic surgery including tumor removal and hip arthroplasty.
  3. presence of bone destruction with soft tissue mass contaminating important organs, nerves and blood vessels (improvement is not expected).
  4. Patients refusing to give a written consent to the study protocol.
  Interventions: Procedure: Percutaneous cementoplasty

INTERVENTIONS:
Procedure: Percutaneous cementoplasty — Percutaneous image guided cementoplasty will be performed as follows:
  Low-viscosity radiopaque bone cement will be quickly mixed and transferred to 1-ml syringes to reduce injection resistance. Injection will be initiated 2-4 min after mixing. When the resistance to cement injection becomes high in the beginning, the cement will be pushed in with a stylet, and it will go well afterward. As much bone cement as possible will be injected while avoiding leakage into the hip joint, sciatic notch, or veins under fluoroscopic monitoring. When significant cement leakage occurred at the initial stage, cement injection will be performed via another route or will be stopped and resumed when the cement viscosity increased. The cement will begin to harden after 8 min, and the operator, therefore, will aim to complete the delivery of the injection within 10 min. The injection needles must be removed before the cement hardens completely

SUMMARY:
This study aimed to summarize the immediate operative and short-term efficacy and safety outcomes of percutaneous cementoplasty for pelvic metastases

DETAILED DESCRIPTION:
Bone metastasis (BM) is the major cause of morbidity in patients with cancer. After lungs and liver, bone is the third most common site of metastatic disease. Prostate and breast cancers are responsible for the majority of bone metastases (up to 70%), followed by thyroid, lung, urinary bladder, and renal cancers, and finally melanoma. The incidence of bone metastasis is approximately 100,000 new cases per year in the united states and is increasing. Bone metastasis could result in skeletal-related events, including pain, pathological fracture, hypercalcemia, and nerve and visceral compression, which seriously affect the quality of life (QoL) of cancer patients. Bone metastases can be classified as osteolytic (osteoclast-mediated bone resorption), osteoblastic (osteoblast-mediated bone deposition), or mixed.

Fifty percent of the pain symptoms experienced by patients with cancer originate from BM. Tumor extension to neural structures, can cause a pain that may be radicular (exacerbated by percussion or palpation) and/or mechanical (exacerbated by movement). In advanced cases, pain can become intolerable and refractory to conventional therapies, resulting in walking disability, psychological and functional impact, and significant worsening of the QoL.

The effectiveness of surgery for bone metastasis in advanced cancer patients is limited to improvement of patients' quality of life. In most of these patients, complete resection or extended curettage of the bone metastasis with major reconstruction is often not feasible due to their poor general condition and accompanying other metastases. For some types of these bone metastases, surgical resection can lead to the stripping of the surrounding soft tissue and muscle attachment and addressing bone defects, causing more intraoperative bleeding, prolonged healing time, and increase the risk of wound complications, which in turn result in a longer recovery time for patients who usually have a limited life expectancy. Therefore, less invasive procedures, including percutaneous ablation (microwave ablation, radiofrequency ablation, cryoablation, and high-energy ultrasound) and/or bone cement [polymethylmethacrylate (PMMA)] injection, have become possible options. This is especially true for pelvic metastatic lesions because the surgery is particularly burdensome.

In addition, life expectancy of patients with metastatic bone disease is the most important factor in the decision making for surgical and/or medical treatment. A short life expectancy is in favor of the use of less invasive procedures, that have lower complication rates and shorter rehabilitation times. In these situations, interventional radiology procedures play an important either primary or complementary role in the management of bone metastases, especially in terms of palliation of pain, improvement of ambulation problems and treatment of fractures. This is because short life expectancies, more often, require palliative rather than curative regimens and make rapid pain relief to become a priority.

Aim of the study This study aimed to summarize the immediate operative and short-term efficacy and safety outcomes of percutaneous cementoplasty for pelvic metastases.

Materials and methods

Target Patients:

The study will include 20 patients with advanced cancer fulfilling the inclusion criteria and giving an informed consent to the study protocol (a single arm).

The following data will be collected from all patients:

1. Age at the time of the procedure
2. Gender
3. Primary cancer
4. Presence of lung metastasis
5. Presence of peritoneal metastasis
6. From the total bone scan:

   1. Unilateral or bilateral pelvic bone metastasis
   2. Solitary or oligometastasis (less than three sites) or multimetastasis ( 3 sites or more).
   3. Presence or absence of spine metastasis
   4. Presence or absence of lower limb metastasis
7. Previous surgery for cancer (site of the operation; pelviabdominal, lower limbs, spine, chest, brain)
8. Chemotherapy (preoperative, postoperative or both)
9. Radiotherapy (preoperative, postoperative or both)

Procedure:

The procedure will be performed under either spinal or general anesthesia. The patient will be placed in the lateral decubitus position with the surgical side up. The needle entry point will be adjusted with a fluoroscopic guide near the point 10 cm posterior to the anterior superior iliac spine. The skin and bone will be punctured by a 11-gauge needle. At least 2 or 3 different routes to the lesion will be established, and one needle will remain empty to allow decompression if possible.

The detailed procedure is described in the intervention section below. During the injection of PMMA, the anesthesiologist carefully will monitor the change in blood pressure and pulse rate, given the known toxicity of bone cement. The injected dose will vary according to the number of metastatic sites injected and their sizes.

All patients who has no contraindication to anticoagulation will be given (enoxaparin 40-60 mg per day) from 1 day before the procedure until ambulation was resumed for deep vein thrombosis prophylaxis.

The following procedural data will be collected:

1. Total cement amount
2. Injection needle number
3. Injection site number
4. Injected sites (Iliac bone or crest, acetabulum, ischium, pubic)
5. Duration of the procedure (in minutes)
6. Type of anesthesia used
7. If any other operation is performed concomitantly (nominate).

Outcome measures:

Primary outcome: is pain reduction:

Secondary outcomes: are

I- Gait function:

1. Gait status will be recorded pre and post operative
2. Gate function change II- Complications of the procedure (if more than one complication occurred in the same patient, all complications will be recorded)

A. Local:

1- Extraosseous bone leakage 2- Pathological fracture of the pelvic bones B. Systemic

1. Mortality
2. Pulmonary embolism
3. Bone cement implantation syndrome (BCIS):

Follow-up outcomes: at one month and 3 months

1. Mortality
2. Pain relapse (NRS score)
3. Gait relapse
4. Pathological fracture in the pelvic bones at the treated sites (by bone window CT).

ELIGIBILITY:
Inclusion Criteria:

1. refractory pain and/or gait disturbance caused by pelvic bone metastasis, did not respond to conservative treatment.
2. osteolytic lesion (in predominance) suitable for the pain.
3. limited life expectancy (less than 3 years) or stopping medical treatment

Exclusion Criteria:

There are no absolute contraindications for the procedure; however, the relative contraindications are:

1. patients in poor condition with an expected survival period of less than 3 months.
2. patients with stable course, with long life expectancy (more than 3 years) or those considered candidates for major pelvic surgery including tumor removal and hip arthroplasty.
3. presence of bone destruction with soft tissue mass contaminating important organs, nerves and blood vessels (improvement is not expected).
4. Patients refusing to give a written consent to the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 3 months
  To evaluate pain, the numerical pain score (NRS) will be used. The NRS is an 11-point numerical scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain (Figure 3) and pain is classified as mild pain if 1-4 points (tolerable), moderate if 5-6 points and severe if 7-10 points. NRS has been shown to be particularly reliable especially among patients with low health literacy. The NRS is also simple to score, and can be administered both orally and in written form.

SECONDARY OUTCOMES:
Gait status | 3 months
  Gait status will be recorded pre and post operative: with the following order from better to worse i. Normal ii. Limping iii. Independent with crutch or cane iv. Wheelchair v. Bed-ridden vi. Dead
Gate function change | 3 months
  i. Improved ii. Stable iii. Worsened
Number of participants with extraosseous cement leakage | 3 months
  It is a safety local outcome that reports extraosseous cement leakage (intra-articular "nominate joint", elsewhere)
Number of participants with pathological fracture of the pelvic bones | 3 months
  A safety local outcome that is reported by history and confirmed by CT that could be impending or displaced
Number of participants with mortality | 3 months
  procedure related mortality is considered within 2 weeks of the procedure
Number of participants with pulmonary embolism | 3 months
  (Pulmonary embolism caused by thrombus, fat, tumor emboli, or bone cement will be diagnosed by pulmonary CT with contrast if clinically suspected). For pulmonary embolism, clinical or radiological factors that might be related to its occurrence were collected, including primary cancer type, presence of lung metastasis, injected cement amount and number, local cement leakage during the procedure, pathologic fracture at the site for procedure, and injected route number.
Number of participants with bone cement implantation syndrome (BCIS) | 3 months
  1- defined as hypoxia, hypertension or both, and/or unexpected loss of consciousness occurring around the time of cementation. BCIS will be classified according to severity of symptoms:
  1. grade 1 was moderate hypoxia (SpO2 < 94%) or hypotension (fall in SBP > 20%)
  2. grade 2 was severe hypoxia (sPO2<88%) or hypotension (fall in SBP>40%) or unexpected loss of consciousness
  3. grade 3 was cardiovascular collapse requiring cardiopulmonary resuscitation (CPR).
Number of participants with pathological fracture in the pelvic bones at the treated sites (by bone window CT) | 3 months
  Local efficacy outcome